CLINICAL TRIAL: NCT04821453
Title: Pilot Cross-Over Trial of Neurally Adjusted Ventilatory Assist (NAVA) and Conventional Flow Triggered Mechanical Ventilation (CMV) in Severe Bronchopulmonary Dysplasia (sBPD)
Brief Title: NAVA vs. CMV Crossover in Severe BPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSME recommendation due to recommendations on study redesign.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Rhode Island Hospital (Other); Children's Miracle Network (Other); American Respiratory Care Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19-017175
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Bronchopulmonary Dysplasia; Neurally Adjusted Ventilatory Assist; Mechanical Ventilation
Keywords: BPD; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Intervention Model Description: Prospective, unblinded, pilot randomized cross-over trial of 2 modes of mechanical ventilation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional Flow Triggered Mechanical Ventilation (CMV) (Placebo Comparator): Subjects will be ventilated with conventional mechanical ventilation with data collected for the 5 day time frame to compare to the experimental arm
  Interventions: Device: CMV
- Neurally Adjusted Ventilatory Assist (NAVA) (Experimental): Subjects will be ventilated on neurally adjusted ventilatory assist (NAVA) mode with data collected for the 5 day time frame to compare with placebo arm
  Interventions: Device: NAVA

INTERVENTIONS:
Device: NAVA — NAVA mode of mechanical ventilation provide the trigger for a spontaneous breath from the diaphragmatic movement instead of diaphragm and allows the patient to control the dynamics of the breath generally set in CMV mode.
  Other Names: Neurally Adjusted Ventilatory Assist
  Arms: Neurally Adjusted Ventilatory Assist (NAVA)
Device: CMV — CMV mode of mechanical ventilation that provides a trigger for a spontaneous breath from the airway flow sensor with dynamics of the breath set as required by the mode
  Other Names: Conventional Flow Triggered Mechanical Ventilation
  Arms: Conventional Flow Triggered Mechanical Ventilation (CMV)

SUMMARY:
This prospective, unblinded, pilot randomized cross-over trial of 2 modes of mechanical ventilation will compare measures of pulmonary mechanics, respiratory gas exchange, and patient comfort between conventional flow triggered mechanical ventilation and neurally adjusted ventilatory assist (NAVA) among 20 prematurely born infants and young children receiving invasive respiratory support for severe bronchopulmonary dysplasia (BPD).

DETAILED DESCRIPTION:
Most research to date in neonatal lung disease has focused on bronchopulmonary dysplasia (BPD) prevention. As a result, insufficient investigation has been performed to define optimal respiratory management strategies for infants and young children with established BPD. Thus, there is no robust evidence base to guide ventilator management to promote lung disease recovery and support neurodevelopment in this population. Neurally adjusted ventilatory assist (NAVA) is an alternative to conventional flow triggered ventilation that has shown promise for improving respiratory gas exchange, patient-ventilator interaction, and work of breathing in preterm neonates. The safety and efficacy of NAVA in infants and young children with established, severe BPD is uncertain. This prospective, unblinded, pilot randomized cross-over trial of 2 modes of mechanical ventilation will compare measures of pulmonary mechanics, respiratory gas exchange, and patient comfort between conventional flow triggered mechanical ventilation and NAVA among 20 prematurely born infants and young children receiving invasive respiratory support for severe BPD.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational ages (GA) ≤ 32 weeks
2. Current age between 36 weeks postmenstrual age (PMA) and 2 years corrected age
3. Severe BPD [as per National Institutes of Health (NIH) consensus definition] diagnosed at 36 weeks postmenstrual age
4. Receiving invasive mechanical ventilation for ongoing lung disease
5. Not expected to be ready for extubation within 11 days following enrollment
6. Parental consent

Exclusion Criteria:

1. Severe congenital anomalies
2. Known diaphragmatic defect
3. Current treatment with high frequency mechanical ventilation
4. Do not resuscitate (DNR) Status or Futility of Care
5. >10% leak around the artificial airway,
6. Treatment with neuromuscular blockade within 72 hours prior to enrollment
7. Acute respiratory instability defined as a ventilator rate increase > 15 beats per minute (bpm), Positive end-expiratory pressure (PEEP) increase > 2 cm/water (H2O), sustained FiO2 increase > 20%, and/or prescribed increase in tidal volume > 2 mL/kg within 24 hours prior to enrollment will be excluded.

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Jensen, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital (Hasboro Children's Hospital), Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 subjects were enrolled in the study and 9 completed the study.
Groups:
- Neurally Adjusted Ventilatory Assist (NAVA) Followed by CMV: Subjects will be ventilated on neurally adjusted ventilatory assist (NAVA) mode with data collected for the first 5 day time, followed by a second day time frame in which subjects will be ventilated with conventional mechanical ventilation (CMV). Data will be collected throughout the two 5 day periods for comaprison.
  NAVA: NAVA mode of mechanical ventilation provide the trigger for a spontaneous breath from the diaphragmatic movement instead of diaphragm and allows the patient to control the dynamics of the breath generally set in CMV mode.
  CMV: CMV mode of mechanical ventilation that provides a trigger for a spontaneous breath from the airway flow sensor with dynamics of the breath set as required by the mode
- Conventional Flow Triggered Mechanical Ventilation (CMV) Followed by NAVA: Subjects will be ventilated with Conventional Mechanical Ventilation (CMV) with for the first 5 day time frame, followed by a second 5 day time frame in which subjects will be ventilated with Neurally Adjusted Ventilatory Assist (NAVA) mode. Data will be collected throughout both 5 day time frames for comparison.
  CMV: CMV mode of mechanical ventilation that provides a trigger for a spontaneous breath from the airway flow sensor with dynamics of the breath set as required by the mode
  NAVA: NAVA mode of mechanical ventilation provide the trigger for a spontaneous breath from the diaphragmatic movement instead of diaphragm and allows the patient to control the dynamics of the breath generally set in CMV mode.
Period: Mechanical Ventilation Sequence 1
Arm/Group | Neurally Adjusted Ventilatory Assist (NAVA) Followed by CMV | Conventional Flow Triggered Mechanical Ventilation (CMV) Followed by NAVA
Started | 7 | 5
Completed | 5 | 5
Not Completed | 2 | 0
Not completed — Unable to complete due to change in patient status. | 1 | 0
Not completed — Patient transferred | 1 | 0
Period: Mechanical Ventilation Sequence 2
Arm/Group | Neurally Adjusted Ventilatory Assist (NAVA) Followed by CMV | Conventional Flow Triggered Mechanical Ventilation (CMV) Followed by NAVA
Started | 5 | 5
Completed | 5 | 4
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: 12 patients were enrolled. 9 completed the study. This is a crossover study design; therefore, each subject completed both arms of the study.
Groups:
- All Study Participants: All study participants include Conventional Flow Triggered Mechanical Ventilation (CMV) and Neurally Adjusted Ventilatory Assist (NAVA)
  CMV: CMV mode of mechanical ventilation that provides a trigger for a spontaneous breath from the airway flow sensor with dynamics of the breath set as required by the mode
  NAVA: NAVA mode of mechanical ventilation provide the trigger for a spontaneous breath from the diaphragmatic movement instead of diaphragm and allows the patient to control the dynamics of the breath generally set in CMV mode.
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Customized [Count of Participants; unit: Participants]
  Under 13 months of age | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Gestational Age at Birth [Number; unit: Count of Participants]
  23-25 weeks | 6
  26-29 weeks | 6
Birth Weight [Number; unit: Count of Participants]
  300-1000 g | 11
  >1000 g | 1

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Saturation (SpO2) Index
Description: The Oxygenation Saturation Index (OSI) is a composite measure of the severity of hypoxic respiratory failure. It quantifies how much ventilatory support is required to achieve a given level of oxygen saturation. Lower OSI values indicate better oxygenation and better clinical status. Higher OSI values indicate worse oxygenation and more severe respiratory failure. Oxygen saturation index will be measured by assessing if invasive mechanical ventilation with NAVA compared to CMV improves respiratory gas exchange in patients receiving invasive respiratory support for BPD. This will be calculated as the mean, time-weighted daily oxygen saturation (SpO2) index ([mean airway pressure x Fraction of inspired oxygen (FiO2)]/SpO2).
Time Frame: up to 5 days per study arm
Population: Three were withdrawn early during the NAVA arm. 2 due to concern for increased hypoxemic episodes and 1 was removed for ventilator technical fault unrelated to patient safety. There is partial data for the 3 subjects who were withdrawn early from the NAVA arm. 1 was never able to be successfully placed on NAVA mode for disordered breathing.
Measure: Mean (Standard Deviation); unit: Oxygen Saturation Index (OSI)
Groups:
- Conventional Mechanical Ventilation (CMV): Subjects will be ventilated with Conventional Mechanical Ventilation (CMV) with data collected for the first 5 day time frame, followed by a second 5 day time frame to compare to the experimental arm.
  CMV: CMV mode of mechanical ventilation that provides a trigger for a spontaneous breath from the airway flow sensor with dynamics of the breath set as required by the mode
- Neurally Adjusted Ventilatory Assist (NAVA): Subjects will be ventilated on neurally adjusted ventilatory assist (NAVA) mode with data collected for the first 5 day time frame, followed by a second 5 day time frame to compare to the experimental arm.
  NAVA: NAVA mode of mechanical ventilation provide the trigger for a spontaneous breath from the diaphragmatic movement instead of diaphragm and allows the patient to control the dynamics of the breath generally set in CMV mode.
Arm/Group | Conventional Mechanical Ventilation (CMV) | Neurally Adjusted Ventilatory Assist (NAVA)
Number analyzed (Participants) | 10 | 9
Oxygen Saturation Index (OSI) | 7.7 (4.7) | 7.7 (4.8)

2. Secondary Outcome: Sedation Medications
Description: The need for sedation medication will be assessed by comparing the needs for sedation by the total daily dose milligram/kilogram (mg/kg) of sedation medications on invasive mechanical ventilation with NAVA compared to CMV.
Time Frame: up to 5 days per study arm
Reporting Status: Not Posted

3. Secondary Outcome: Stress
Description: Patient stress will be assessed by collecting salivary swabs three times per day to measure cortisol levels. The daily average will be assessed and compared as a marker for patient stress on invasive mechanical ventilation with NAVA compared to CMV.
Time Frame: up to 5 days per study arm
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 11 days
Description: Due to the medical complexity of subjects, only intervention related AEs were captured.
Arm/Group | Conventional Flow Triggered Mechanical Ventilation (CMV) | Neurally Adjusted Ventilatory Assist (NAVA)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Flow Triggered Mechanical Ventilation (CMV) (N=12) | Neurally Adjusted Ventilatory Assist (NAVA) (N=12)
Increased risk for Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (18) — concern for increased hypoxemic episodes
Procedural Event (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Vaso-vagal response with insertion of NAVA catheter

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT04821453/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT04821453/ICF_001.pdf